CLINICAL TRIAL: NCT03818074
Title: A Prospective Single Centre Pilot Study to Investigate the Response to 1000Hz Frequency in Patients With Spinal Cord Stimulation With Intractable Neuropathic Pain Who Have Not Undergone Spinal Surgery (Virgin Back)
Brief Title: High Frequency (1000Hz) Spinal Cord Stimulation in Neuropathic Pain Patients With Virgin Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012170
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Neuropathic Pain; Low Back Pain
Keywords: High Frequency spinal cord stimulation
MeSH Terms: conditions — Neuralgia; Low Back Pain

STUDY DESIGN:
Intervention Model Description: To investigate the clinical response to high frequency (1,000Hz) in patients who are due to have percutaneous spinal cord stimulation for intractable back and lower limb neuropathic pain
Masking Description: Patients will be required to adhere to the study and attend all follow up visits. Informed consent and questionnaires will be administered at visit 0. They will be followed up 4, 12, 24 weeks and 12 months, 24 months after their SCS permanent implant. Questionnaires will be administered at each visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Boston Wavewriter (1000Hz) spinal cord stimulation (Experimental): To investigate the response to high frequency (1000Hz) in patients who are due to have spinal cord stimulation for neuropathic back pain.
  Interventions: Device: Boston Wavewriter 1000Hz Spinal cord Stimulation

INTERVENTIONS:
Device: Boston Wavewriter 1000Hz Spinal cord Stimulation — High frequency spinal cord stimulation.

SUMMARY:
Spinal Cord stimulation (SCS) is a common intervention used in patients who suffer from chronic nerve pain following back surgery. This is known as failed back surgery syndrome (FBSS). Equally, the National Institute of Clinical Excellence (NICE) who work with the NHS, recommend suitable medicines and treatments for patients in their guidelines; suggest that SCS can be used in patients who have never had back surgery. The is no outcome data to define that SCS works in patients with neuropathic back pain, therefore this study will provide clinical data to see if this works.

SCS delivers mild electrical impulses to the nerves along the spinal cord. This blocks the pain pathway from reaching the brain. This helps manage the pain experienced the lower back.

A common side effect of the conventional system is that patients may experience 'pins and needles', tingling, and numbness, known as parathesia at site of stimulation. This can be particularly uncomfortable for patients. However, parathesia can be eliminated by changing certain settings on the stimulator. This could include increasing the frequency of the stimulator known as high frequency (HF). This works by delivering energy to site of stimulation below the parathesia threshold, so minimal or no parathesia is experienced.

Only one study has been completed previously using HF frequency on patients with FBSS. The major findings from these studies have found that when compared to conventional SCS (uses a frequency of 40-80 Hz) that HF has provided better pain relief with minimal or no parathesia. Higher frequencies parameters are not completely novel because they have been used in patients who have FBSS. However, settings of 1000Hz which will be used in this study have not been done in patients who suffer from neuropathic pain and have not had any previous spinal surgery.

Therefore, the main reason of this study is to investigate the response patients suffering from neuropathic pain and have not had previous spinal surgery, have to 1000Hz (HF) frequency spinal cord stimulation. We will also investigate the effect this setting has on the quality of life of the patients.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) is a successful treatment in patients with intractable neuropathic pain. This therapy is most commonly used in patients who have chronic neuropathic pain following failed surgery, known as failed back surgery syndrome (FBSS) . There is evidence from previous studies to demonstrate that SCS can provide a 50- 70% reduction in pain medication and pain scores. A randomised controlled study compared SCS with conventional medical management (CMM). When compared with the CMM group; the SCS patients had a 50% pain reduction in their back pain and leg pain. The results suggested that patients who received SCS had better pain relief and health related quality of life over a period of 6 to 12 months compared to the CMM group. Additionally, these patients reported satisfaction in SCS treatment, continuous pain relief, and clinical improvements in functional capacity and health-related quality of life.

On the other hand, SCS has been progressively being used in patients with intractable neuropathic pain who have not undergone spinal back surgery ("Virgin-back''). The UK NICE guidelines have recommended SCS as a treatment option for patients with intractable neuropathic spinal pain, including patients who have not undergone previous spinal surgery (NICE, 2008).

One of the main drawbacks of conventional SCS is the onset of parathesia, despite being an effective therapy for neuropathic pain. This can cause abnormal sensations or considerable discomfort to the patient during activity or sudden position changes. Typically, conventional SCS operate at frequencies ranging from 40-80 Hz, long pulse widths of 300-500 µsec, and amplitudes to stimulate patient's pain sensory percept distribution. These frequencies are often used because sensory perception is often lost at 300 Hz. Current studies have found that delivering stimulating frequencies below the upper limit of what may cause parathesia; may reduce discomfort and abnormal sensations, increasing the tolerability of SCS treatment. Parathesia is considered necessary in order to cover the painful area and provide maximum pain relief. However recent research suggests that parathesia may not be necessary for pain relief, and in fact that pain awareness can provide full benefits of SCS.

Data from (PROCO RCT) indicates that similar pain relief and improvement in quality of life measures are experienced independent of the type of frequency (from 1kHz up to 10kHz) used in paraesthesia free SCS therapy when the proper target and dose are identified. Further, the study showed that 1kHz stimulation provides similar pain relief using significantly less energy than higher frequencies.

High frequency (HF) stimulation is a new promising, new stimulation paradigm involving higher frequency, lower pulse widths, and lower amplitudes when compared to conventional SCS. The effectiveness of HF-SCS is controlled by the amount of Neural dose (frequency, amplitude and pulse width) passing the electrodes and reaching the neural tissue, resulting in minimal discomfort and damage to the tissues before the definite shape of the impulse.

Pre-clinical Data

A study testing the efficacy of kilohertz and conventional SCS was done on rat models during different pain conditions. The findings established that higher frequencies can be delivered at lower amplitudes whilst reversing pain behaviours as seen at 50 Hz and at higher intensity of motor threshold.

Moreover, both conventional and kilohertz frequency SCS forms intensity and frequency-dependant inhibition of mechanical hypersensitivity, in animal models of neuropathic pain. Different intensities (20, 40 and 80% motor threshold) and frequencies (50, 1kHz and 10kHz) were used. At each frequency, the pulse width was constant. It was observed that as frequency was increased, the pulse density also increased.

Clinical data

Previous randomised control trials have provided evidence that using frequency ≤1200 Hz and pulses ≤ 5% provides efficient relief with HF- SCS.

A multi-centre trial previously conducted to see the effects of HF-SCS on patients being delivered up to 10 kHz of stimulation. Patients were assessed for pain ratings, disability, sleep disturbances, and satisfaction, as well as complication rates for up to six months. When results were compared to baseline, 88% of patients reported a significant reduction in mean back visual analogue scores (VAS) from 8.4 to 2.7 at six months. Seventy four per cent of patients reported more than 50% back pain relief at six months. Overall it was concluded that individuals in the trial group with chronic back pain, 70% of patients were provided with positive improvement and experienced sustained low back and leg pain relief. Substantial improvements were also seen for these patients with disability and sleep disturbances.

If clinically considered, the NRS has substantially reduced in patients who received HF-SCS than conventional SCS in patients with neuropathic pain and FBSS. This suggests that HF may provide relief in virgin-back patients. Since there remains limited research in this area therefore, the main objective of our study is to investigate the response to 1000Hz frequency following SCS treatment in "virgin back" patients with intractable lower limb neuropathic pain. However based on the PROCO RCT and further WHISPER trial, we aim to establish role of microburst and combination therapy in non-responders.

Our sample size of 30 patients will allow detection of minimal important difference of 2.0 on the NRS pain scale at 90% power and alpha of 5%, assuming an outcome standard deviation of 2.5 and attrition rate at 12-months of 30%. Patient primary and secondary outcomes at each follow up point will be compared to baseline values. Data analyses will take account of the paired nature of the data and use non-independent t-test for continuous outcomes and McNemar's test for binary outcomes.

* The primary objective is to investigate the clinical response to high frequency (1,000Hz) in patients who are due to have percutaneous spinal cord stimulation for intractable lower limb neuropathic pain
* The secondary objective will be to investigate the effect on functionality and quality of life and adverse events at the high frequency group (1000Hz)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70
2. Chronic Back Pain (≥ 6 mo) with NRS ≥ 6/10
3. Back pain predominant over leg pain (if leg pain present)
4. Failure to respond to conventional treatment including intense rehababilitation and facet/MBB/SI interventions
5. No prior spinal surgery for the back and leg pain on the same site of implantation.
6. Presence of lumbar degenerative disc disease
7. Absence of spinal pathology which would require surgical intervention
8. Stable dose of opioids and anti-neuropathic drugs for ≥ 6 months
9. Patients with intractable lumbar neuropathic pain who are due to receive Percutaneous Spinal Cord Stimulation as part of their standard treatment per NICE HTA guidance 159 at Barts Health NHS Hospitals.
10. Patients who have given their written informed consent.
11. Female patients of childbearing potential must be using adequate contraception (i.e. using oral or IM contraception or an IUCD) and must have a negative urine pregnancy test.
12. Patients must be able to communicate in English in order to complete validated questionnaires written in English.

Exclusion Criteria:

1. Patients not able to comply or understand the study-related requirements
2. Active alcohol, recreational or prescription drug abuse in the last 3 months.
3. Unwilling to reduce excessive pain medications
4. A medical/psychiatric condition that could interfere with study procedures, accurate pain reporting, and/or confound study outcomes
5. Patients with diabetes or any current diagnosis of progressive neurological disease (i.e., CIDP, Multiple sclerosis)
6. Immuno-compromised/high risk for surgical infection
7. Pregnant and/or breast feeding
8. Terminal illness with anticipated survival < 12 months
9. Patients who have been part of a previous spinal cord stimulation trial
10. Currently implanted with an active implantable device(s) (e.g. pacemaker, drug pump, implantable pulse generator)
11. Untreated clinically significant sleep disorder as judged by the CI.
12. Unresolved issues of secondary gain (i.e., litigation)
13. Participation in another clinical study in the last 30 days that would confound data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline numerical Rating Score (NRS) at 4 weeks | 4 weeks
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale. An average overall pain score will be recorded over the last 7 days.
change from baseline numerical Rating Score (NRS) at 3 months | 3 months
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale. An average overall pain score will be recorded over the last 7 days.
Change from baseline numerical Rating Score (NRS) at 6 months | 6 months
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale. An average overall pain score will be recorded over the last 7 days.
Change from baseline numerical Rating Score (NRS) at 12 months | 12 months
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale. An average overall pain score will be recorded over the last 7 days.
Change from baseline numerical Rating Score (NRS) at 24 months | 24 months
  NRS will be used to measure the pain intensity, enabling the patient to express the severity of pain by giving it a numerical value from 0 to 10 on an 11-point numerical pain rating scale. An average overall pain score will be recorded over the last 7 days.
Change from baseline Oswestry Disability Index (ODI) scores at 4 weeks | 4 weeks
  A commonly used scale for back pain patients with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Change from baseline Oswestry Disability Index (ODI) scores at 3 months | 3 months
  A commonly used scale for back pain patients with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Change from baseline Oswestry Disability Index (ODI) scores at 6 months | 6 months
  A commonly used scale for back pain patients with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Change from baseline Oswestry Disability Index (ODI) scores at 12 months | 12 months
  A commonly used scale for back pain patients with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Change from baseline Oswestry Disability Index (ODI) scores at 24 months | 24 months
  A commonly used scale for back pain patients with a neuropathic pain component. The test is considered the 'gold standard' of low back functional outcome tools.
Change from baseline Patient's Global Impression of change (PGIC) scores to 4 weeks | 4 weeks
  A standard seven point scale would be used to assess the SCS outcome.
Change from baseline Patient's Global Impression of change (PGIC) scores to 3 months | 3 months
  A standard seven point scale would be used to assess the SCS outcome.
Change from baseline Patient's Global Impression of change (PGIC) scores to 6 months | 6 months
  A standard seven point scale would be used to assess the SCS outcome.
Change from baseline Patient's Global Impression of change (PGIC) scores to 12 months | 12 months
  A standard seven point scale would be used to assess the SCS outcome.
Change from baseline Patient's Global Impression of change (PGIC) scores to 24 months | 24 months
  A standard seven point scale would be used to assess the SCS outcome.
change from baseline EQ-5D-5L scores at 4 weeks | 4 weeks
  The EQ-5D is a standardised instrument used to measure health outcome.
change from baseline EQ-5D-5L scores at 3 months | 3 months.
  The EQ-5D is a standardised instrument used to measure health outcome.
change from baseline EQ-5D-5L scores at 6 months | 6 months.
  The EQ-5D is a standardised instrument used to measure health outcome.
change from baseline EQ-5D-5L scores at 12 months | 12 months.
  The EQ-5D is a standardised instrument used to measure health outcome.
change from baseline EQ-5D-5L scores at 24 months | 24 months.
  The EQ-5D is a standardised instrument used to measure health outcome.
Change from baseline Pain and Sleep 3 point index (PSQ-3) at 4 weeks | 4 weeks
  The PSQ-3 is an instrument that measures the quality of sleep over a month.
Change from baseline Pain and Sleep 3 point index (PSQ-3) at 3 months | 3 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month.
Change from baseline Pain and Sleep 3 point index (PSQ-3) at 6 months | 6 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month.
Change from baseline Pain and Sleep 3 point index (PSQ-3) at 12 months | 12 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month.
Change from baseline Pain and Sleep 3 point index (PSQ-3) at 24 months | 24 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month.
Change from baseline Resource Questionnaire at 12 months | 12 months.
  The resource questionnaire measures the impact of health on employment.
Change from baseline Resource Questionnaire at 24 months | 24 months.
  The resource questionnaire measures the impact of health on employment.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Poply, Dr, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Vivek Health Mehta, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will follow the policies laid by the local information governance team at Barts Health NHS Trust and NHS code of Confidentiality in accordance to the data protection act.